CLINICAL TRIAL: NCT00106028
Title: Safety and Efficacy of Risedronate in the Treatment of Osteogenesis Imperfecta in Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Warner Chilcott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2003100; HMR4003I/3001
Record Dates: First submitted 2005-03-18; First posted 2005-03-21 (Estimated); Results first posted 2010-06-28 (Estimated); Last update posted 2013-04-22 (Estimated); Status verified 2013-04

CONDITIONS: Osteogenesis Imperfecta
Keywords: Primary disease: Osteogenesis Imperfecta
MeSH Terms: conditions — Osteogenesis Imperfecta | interventions — Risedronic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo Daily (Placebo Comparator): placebo tablet, once a day for one year then for two years open label risedronate
  Interventions: Drug: Placebo
- Risedronate Daily (Experimental): risedronate tablet, once a day for one year then for two years open label risedronate once a day
  Interventions: Drug: risedronate sodium (Actonel)

INTERVENTIONS:
Drug: risedronate sodium (Actonel) — risedronate tablet once a day for one year followed by risedronate once a day for two years
  Arms: Risedronate Daily
Drug: Placebo — placebo tablet once a day for one year followed by risedronate once a day for two years
  Arms: Placebo Daily

SUMMARY:
Children with Osteogenesis Imperfecta (OI) have bone pain, low bone mass and fractures. There are no approved drugs for the treatment of OI in children, even though some intravenous (IV) bisphosphonates are used off-label in some countries. In a single dose, pharmacokinetic study, data showed that risedronate was well tolerated in 28 children with OI. This three year study will test the safety and efficacy of risedronate in the treatment of children with OI. For the first year, patients will be randomized to the risedronate and placebo groups in a 2:1 ratio. For the second and third years of the study, all patients will receive risedronate.

ELIGIBILITY:
Inclusion Criteria:

* OI diagnosis
* increased risk of fracture: either has a history of at least 1 radiographically confirmed, non-traumatic or low impact fracture plus low bone mineral density (BMD) or has very low BMD with or without a history of fractures.

Exclusion Criteria:

* Any bisphosphonate use within one year of enrollment

Ages: 4 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 143 (Actual)
Dates: Start 2004-11; Primary Completion 2008-04 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dietrich H Wenderoth, MD, Study Director — Procter and Gamble
Locations (20):
- United States (5):
  - Miami Children's Hospital, Miami, Florida
  - University of Nebraska Medical Center, Children's Hospital, Omaha, Nebraska
  - Hospital for Special Surgery, New York, New York
  - Wright State University BioMedical Imaging Laboratory and Miami Valley Hospital, Dayton, Ohio
  - Oregon Health & Science University, Portland, Oregon
- Australia (2):
  - The Children's Hospital at Westmead, Westmead, New South Wales
  - Princess Margaret Hospital for Children, Perth
- Cliniques Universitaires Saint Luc, Brussels, Belgium
- Pontificia Universidad Catolica de Chile, Santiago, Chile
- Osteocentrum, II. Interní klinika, Fakultní nemocnice Plzeň-Bory, Pilsen, Czechia
- Hospital for Children and Adolescents, Helsinki, Finland
- Klinikum und Poliklinik für Kinderheilkunde der Universität zu Köln, Cologne, Germany
- 2nd Department of Pediatrics, Semmelwies University, Faculty of Medicine, Budapest, Hungary
- Rheumatologic Rehabilitation Unit of the University of Verona, Valeggio sul Mincio, Italy
- Zaklad Biochemii i Medycyny Doswiadczalnej (Biochemisty Dept, Institute "Monument-Children Health Centre", Warzawa-Międzylesie, Poland
- Little Company of Mary Hospital, Pretoria, Gauteng, South Africa
- Hospital Sant Joan de Deu, Barcelona, Spain
- United Kingdom (3):
  - Royal Hospital for Sick Children, Glasgow, Glasgow
  - Sheffield Children's Hospital, Sheffield, Sheffield
  - Bristol Royal Hospital for Children,, Bristol

REFERENCES:
- [Derived] Bishop N, Adami S, Ahmed SF, Anton J, Arundel P, Burren CP, Devogelaer JP, Hangartner T, Hosszu E, Lane JM, Lorenc R, Makitie O, Munns CF, Paredes A, Pavlov H, Plotkin H, Raggio CL, Reyes ML, Schoenau E, Semler O, Sillence DO, Steiner RD. Risedronate in children with osteogenesis imperfecta: a randomised, double-blind, placebo-controlled trial. Lancet. 2013 Oct 26;382(9902):1424-32. doi: 10.1016/S0140-6736(13)61091-0. Epub 2013 Aug 6. PMID 23927913

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 147 children > or = 4 and < 16 years of age with Osteogenesis Imperfecta (OI) enrolled at 20 North American and international study centers starting 16NOV2004. Patients weighing 10-30 kg received risedronate 2.5 mg or placebo daily and patients weighing more than 30 kg received risedronate 5 mg or placebo daily.
Period: Overall Study
Arm/Group | Placebo Daily | Risedronate Daily
Started | 49 (ITT Population: Patients Randomized and Received at least 1 Dose of Study Drug) | 94 (ITT Population: Patients Randomized and Received at least 1 Dose of Study Drug)
Month 12 Completed/Started Open Label | 49 | 87
Completed | 43 (Completed Month 36) | 82 (Completed Month 36)
Not Completed | 6 | 12
Not completed — Adverse Event | 3 | 2
Not completed — Protocol Violation | 1 | 1
Not completed — Withdrawal by Subject | 2 | 8
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Daily | Risedronate Daily | Total
Number analyzed (Participants) | 49 | 94 | 143
Age, Categorical [Count of Participants; unit: Participants] — There were 147 children enrolled in the study (stated in the protocol). However, 4 children were randomized but did not receive a dose of the study drug. Therefore, only 143 received at least 1 dose of study drug.
  Participants
    <=18 years | 49 | 94 | 143.0
    Between 18 and 65 years | 0 | 0 | 0.0
    >=65 years | 0 | 0 | 0.0
Age Continuous [Mean (Standard Deviation); unit: years] | 8.6 (3.1) | 8.9 (3.4) | 8.825 (3.313)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 49 | 71.0
  Male | 27 | 45 | 72.0
Region of Enrollment [Number; unit: participants]
  Australia | 8 | 16 | 24.0
  Belgium | 1 | 1 | 2.0
  Chile | 4 | 9 | 13.0
  Czech Republic | 1 | 4 | 5.0
  Finland | 5 | 7 | 12.0
  Germany | 5 | 8 | 13.0
  Hungary | 2 | 2 | 4.0
  Italy | 1 | 2 | 3.0
  Poland | 5 | 9 | 14.0
  South Africa | 0 | 1 | 1.0
  Spain | 1 | 1 | 2.0
  United Kingdom | 9 | 21 | 30.0
  United States | 7 | 13 | 20.0

OUTCOME MEASURES:

1. Secondary Outcome: Percent Change From Baseline Lumbar Spine Bone Mineral Density (BMD) at Month 24, ITT Population
Description: Lumbar Spine Bone Mineral Density (BMD) measured by dual-energy x-ray absorptiometry (DXA)and read by central reader.
Time Frame: Baseline and Month 24
Population: ITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Placebo Daily | Risedronate Daily
Number analyzed (Participants) | 49 | 94
Percent Change | 21.316 [17.357 to 25.275] | 25.754 [22.860 to 28.648]
Statistical Analysis 1: Comparison: Placebo Daily vs Risedronate Daily; A total of 123 patients were to be randomized in 2:1 ratio. The sample size allowed detection of a difference of at least 5% in lumbar spine BMD percent change from baseline to 12 months with 90% power. Calculation based on assumption that common within-group SD would be approximately 7% and dropout rate within Year 1 would be 20%. A difference of 5% in lumbar spin BMD percent change from baseline was considered clinically meaningful; Test type: Superiority or Other; p = 0.0625, ANCOVA; LS means and p-value are from ANCOVA model adjusted by baseline and fixed effects for age group, treatment and pooled center for post-baseline; Mean Difference (Net) = 4.438, 95% CI 2-sided [-0.235 to 9.111]

2. Secondary Outcome: Percent Change From Baseline Lumbar Spine Bone Mineral Density (BMD) at Month 36, ITT Population
Description: Lumbar Spine Bone Mineral Density (BMD) measured by dual-energy x-ray absorptiometry (DXA)and read by central reader.
Time Frame: Baseline and Month 36
Population: ITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Placebo Daily | Risedronate Daily
Number analyzed (Participants) | 49 | 94
Percent Change | 33.216 [28.191 to 38.241] | 34.753 [31.076 to 38.429]
Statistical Analysis 1: Comparison: Placebo Daily vs Risedronate Daily; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.6103, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 1.537, 95% CI 2-sided [-4.424 to 7.497]

3. Secondary Outcome: Percent Change From Baseline in Total Body BMD at Month 12, ITT Population
Description: Percent Change from baseline in Total Body Bone Mineral Density (BMD) measured by DXA.
Time Frame: Baseline and Month 12
Population: ITT Population.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Placebo Daily | Risedronate Daily
Number analyzed (Participants) | 49 | 94
Percent Change | 4.252 [2.762 to 5.743] | 5.806 [4.740 to 6.872]
Statistical Analysis 1: Comparison: Placebo Daily vs Risedronate Daily; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0808, ANCOVA; LS means and p-value are from ANCOVA model adjusted by baseline and with fixed effects for age group, treatment and pooled center for post-baseline; Mean Difference (Net) = 1.554, 95% CI [-0.193 to 3.301]

4. Secondary Outcome: Percent Change From Baseline in Total Body BMD at Month 24, ITT Population
Description: Percent Change from baseline in Total Body Bone Mineral Density (BMD) measured by DXA.
Time Frame: Baseline and Month 24
Population: ITT Population.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Placebo Daily | Risedronate Daily
Number analyzed (Participants) | 49 | 94
Percent Change | 9.716 [7.897 to 11.535] | 10.214 [8.899 to 11.528]
Statistical Analysis 1: Comparison: Placebo Daily vs Risedronate Daily; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.6466, ANCOVA; [statistical method as in outcome 3, analysis 1]; Mean Difference (Net) = 0.498, 95% CI 2-sided [-1.648 to 2.644]

5. Secondary Outcome: Percent Change From Baseline in Total Body BMD at Month 36, ITT Population
Description: Percent Change from baseline in Total Body Bone Mineral Density (BMD) measured by DXA.
Time Frame: Baseline and Month 36
Population: ITT Population.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Placebo Daily | Risedronate Daily
Number analyzed (Participants) | 49 | 94
Percent Change | 13.540 [11.204 to 15.876] | 13.076 [11.374 to 14.777]
Statistical Analysis 1: Comparison: Placebo Daily vs Risedronate Daily; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.7391, ANCOVA; [statistical method as in outcome 3, analysis 1]; Mean Difference (Net) = -0.465, 95% CI 2-sided [-3.224 to 2.294]

6. Secondary Outcome: Percent Change From Baseline in Lumbar Spine BMC (Bone Mineral Content) at Month 12, ITT Population
Time Frame: Baseline and Month 12
Population: ITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Placebo Daily | Risedronate Daily
Number analyzed (Participants) | 49 | 94
Percent Change | 17.885 [13.645 to 22.124] | 28.218 [25.038 to 31.398]
Statistical Analysis 1: Comparison: Placebo Daily vs Risedronate Daily; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 3, analysis 1]; Mean Difference (Net) = 10.333, 95% CI [5.258 to 15.408]

7. Secondary Outcome: Percent Change From Baseline in Lumbar Spine BMC (Bone Mineral Content) at Month 24, ITT Population
Time Frame: Baseline and Month 24
Population: ITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Placebo Daily | Risedronate Daily
Number analyzed (Participants) | 49 | 94
Percent Change | 42.367 [34.871 to 49.863] | 48.407 [42.921 to 53.894]
Statistical Analysis 1: Comparison: Placebo Daily vs Risedronate Daily; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 01789, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 6.040, 95% CI 2-sided [-2.807 to 14.887]

8. Secondary Outcome: Percent Change From Baseline in Lumbar Spine BMC (Bone Mineral Content) at Month 36, ITT Population
Time Frame: Baseline and Month 36
Population: ITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Placebo Daily | Risedronate Daily
Number analyzed (Participants) | 49 | 94
Percent Change | 68.054 [57.564 to 78.544] | 68.333 [60.607 to 76.060]
Statistical Analysis 1: Comparison: Placebo Daily vs Risedronate Daily; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.9646, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.280, 95% CI 2-sided [-12.196 to 12.755]

9. Secondary Outcome: Percent Change From Baseline in Total Body BMC at Month 12, ITT Population
Time Frame: Baseline and Month 12
Population: ITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Placebo Daily | Risedronate Daily
Number analyzed (Participants) | 49 | 94
Percent Change | 16.483 [13.395 to 19.570] | 21.977 [19.772 to 24.181]
Statistical Analysis 1: Comparison: Placebo Daily vs Risedronate Daily; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0030, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 5.494, 95% CI [1.912 to 9.077]

10. Secondary Outcome: Percent Change From Baseline in Total Body BMC at Month 24, ITT Population
Time Frame: Baseline and Month 24
Population: ITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Placebo Daily | Risedronate Daily
Number analyzed (Participants) | 49 | 94
Percent Change | 36.465 [31.582 to 41.347] | 37.938 [34.406 to 41.470]
Statistical Analysis 1: Comparison: Placebo Daily vs Risedronate Daily; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.6106, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 1.473, 95% CI 2-sided [-4.245 to 7.192]

11. Secondary Outcome: Percent Change From Baseline in Total Body BMC at Month 36, ITT Population
Time Frame: Baseline and Month 36
Population: ITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Placebo Daily | Risedronate Daily
Number analyzed (Participants) | 49 | 94
Percent Change | 56.211 [49.470 to 62.952] | 56.526 [51.549 to 61.503]
Statistical Analysis 1: Comparison: Placebo Daily vs Risedronate Daily; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.9372, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.315, 95% CI 2-sided [-7.598 to 8.229]

12. Secondary Outcome: Lumbar Spine Z-score - Percent Change From Baseline to Month 12, ITT Population
Description: Lumbar Spine Z-score - number of standard deviations a patient's BMD differs from the average BMD of their age, sex, and ethnicity. Positive scores indicate BMD above the mean; Positive values are "best values" and negative values are "worst values".
Time Frame: Baseline and Month 12
Population: ITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a Scale
Arm/Group | Placebo Daily | Risedronate Daily
Number analyzed (Participants) | 49 | 94
Units on a Scale | -6.028 [-14.899 to 2.844] | 25.648 [18.993 to 32.302]
Statistical Analysis 1: Comparison: Placebo Daily vs Risedronate Daily; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS means and p-value are from ANCOVA model adjusted for baseline and fixed effects for age group, treatment and pooled center for post-baseline; Mean Difference (Net) = 31.675, 95% CI [21.051 to 42.300]

13. Secondary Outcome: Lumbar Spine Z-score - Percent Change From Baseline to Month 24, ITT Population
Description: as for outcome 12
Time Frame: Baseline and Month 24
Population: ITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a Scale
Arm/Group | Placebo Daily | Risedronate Daily
Number analyzed (Participants) | 49 | 94
Units on a Scale | 15.608 [2.327 to 28.889] | 29.637 [19.911 to 39.363]
Statistical Analysis 1: Comparison: Placebo Daily vs Risedronate Daily; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0793, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 14.029, 95% CI 2-sided [-1.667 to 29.726]

14. Primary Outcome: Percent Change From Baseline Lumbar Spine Bone Mineral Density (BMD) at Month 12, ITT Population
Description: Lumbar Spine Bone Mineral Density (BMD) measured by dual-energy x-ray absorptiometry (DXA)and read by central reader. Duplicate scans obtained at screening and Month 12.
Time Frame: Baseline and Month 12
Population: ITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Placebo Daily | Risedronate Daily
Number analyzed (Participants) | 49 | 94
Percent Change | 7.592 [5.106 to 10.078] | 16.159 [14.295 to 18.024]
Statistical Analysis 1: Comparison: Placebo Daily vs Risedronate Daily; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 3, analysis 1]; Mean Difference (Net) = 8.567, 95% CI [5.590 to 11.545]

15. Secondary Outcome: Lumbar Spine Z-score - Percent Change From Baseline to Month 36, ITT Population
Description: as for outcome 12
Time Frame: Baseline and Month 36
Population: ITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a Scale
Arm/Group | Placebo Daily | Risedronate Daily
Number analyzed (Participants) | 49 | 94
Units on a Scale | 19.325 [5.162 to 33.488] | 25.640 [15.313 to 35.967]
Statistical Analysis 1: Comparison: Placebo Daily vs Risedronate Daily; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.4575, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 6.315, 95% CI 2-sided [-10.477 to 23.107]

16. Secondary Outcome: Total Body Z-score- Percent Change From Baseline to Month 12, ITT Population
Description: Total Body Z-score - number of standard deviations a patient's BMD differs from the average BMD of their age, sex, and ethnicity. Positive scores indicate BMD above the mean; Positive values are "best values" and negative values are "worst values".
Time Frame: Baseline and Month 12
Population: ITT Population, Population Description Number of Participants Analyzed = Number of participants at baseline and LOCF data
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a Scale
Arm/Group | Placebo Daily | Risedronate Daily
Number analyzed (Participants) | 49 | 94
Units on a Scale | -20.661 [-47.090 to 5.769] | 16.933 [-1.793 to 35.660]
Statistical Analysis 1: Comparison: Placebo Daily vs Risedronate Daily; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0172, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 37.594, 95% CI [6.801 to 68.386]

17. Secondary Outcome: Total Body Z-score- Percent Change From Baseline to Month 24, ITT Population
Description: as for outcome 16
Time Frame: Baseline and Month 24
Population: ITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a Scale
Arm/Group | Placebo Daily | Risedronate Daily
Number analyzed (Participants) | 49 | 94
Units on a Scale | 8.371 [-22.631 to 39.373] | 7.879 [-14.273 to 30.032]
Statistical Analysis 1: Comparison: Placebo Daily vs Risedronate Daily; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.9786, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.492, 95% CI 2-sided [-36.807 to 35.824]

18. Secondary Outcome: Total Body Z-score- Percent Change From Baseline to Month 36, ITT Population
Description: as for outcome 16
Time Frame: Baseline and Month 36
Population: ITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a Scale
Arm/Group | Placebo Daily | Risedronate Daily
Number analyzed (Participants) | 49 | 94
Units on a Scale | 7.146 [-20.474 to 34.766] | -1.494 [-21.400 to 18.411]
Statistical Analysis 1: Comparison: Placebo Daily vs Risedronate Daily; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.5971, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -8.640, 95% CI 2-sided [-40.952 to 23.672]

19. Secondary Outcome: Percent Change From Baseline in Lumbar Spine Bone Area at Month 12, ITT Population
Description: Measured by DXA.
Time Frame: Baseline and Month 12
Population: ITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Placebo Daily | Risedronate Daily
Number analyzed (Participants) | 49 | 94
Percent Change | 8.803 [6.751 to 10.856] | 9.817 [8.278 to 11.356]
Statistical Analysis 1: Comparison: Placebo Daily vs Risedronate Daily; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.4154, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 1.014, 95% CI [-1.442 to 3.470]

20. Secondary Outcome: Percent Change From Baseline in Lumbar Spine Bone Area at Month 24, ITT Population
Description: Measured by DXA.
Time Frame: Baseline and Month 24
Population: ITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Placebo Daily | Risedronate Daily
Number analyzed (Participants) | 49 | 94
Percent Change | 16.381 [13.214 to 19.549] | 17.266 [14.945 to 19.586]
Statistical Analysis 1: Comparison: Placebo Daily vs Risedronate Daily; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.6404, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.884, 95% CI 2-sided [-2.855 to 4.623]

21. Secondary Outcome: Percent Change From Baseline in Lumbar Spine Bone Area at Month 36, ITT Population
Description: Measured by DXA.
Time Frame: Baseline and Month 36
Population: ITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Placebo Daily | Risedronate Daily
Number analyzed (Participants) | 49 | 94
Percent Change | 24.952 [20.877 to 29.027] | 23.292 [20.296 to 26.289]
Statistical Analysis 1: Comparison: Placebo Daily vs Risedronate Daily; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.4978, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -1.660, 95% CI 2-sided [-6.499 to 3.179]

22. Secondary Outcome: Percent Change From Baseline in Total Body Bone Area Month 12, ITT Population
Time Frame: Baseline and Month 12
Population: ITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Placebo Daily | Risedronate Daily
Number analyzed (Participants) | 49 | 94
Percent Change | 11.405 [8.708 to 14.101] | 14.939 [13.028 to 16.850]
Statistical Analysis 1: Comparison: Placebo Daily vs Risedronate Daily; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0270, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 3.534, 95% CI [0.410 to 6.658]

23. Secondary Outcome: Percent Change From Baseline in Total Body Bone Area Month 24, ITT Population
Time Frame: Baseline and Month 24
Population: ITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Placebo Daily | Risedronate Daily
Number analyzed (Participants) | 49 | 94
Percent Change | 24.051 [20.684 to 27.417] | 25.116 [22.699 to 27.533]
Statistical Analysis 1: Comparison: Placebo Daily vs Risedronate Daily; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.5925, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 1.065, 95% CI 2-sided [-2.868 to 4.998]

24. Secondary Outcome: Percent Change From Baseline in Total Body Bone Area Month 36, ITT Population
Time Frame: Baseline and Month 36
Population: ITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Placebo Daily | Risedronate Daily
Number analyzed (Participants) | 49 | 94
Percent Change | 37.109 [32.144 to 42.074] | 38.303 [34.674 to 41.931]
Statistical Analysis 1: Comparison: Placebo Daily vs Risedronate Daily; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.6840, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 1.193, 95% CI 2-sided [-4.604 to 6.991]

25. Secondary Outcome: New Morphometric Vertebral Fracture at Month 12, ITT Population
Description: Morphometric Vertebral Fracture measured by semi-quantitative (SQ) analysis of x-rays using the Genant scoring system at endpoint. (Ref: Genant 1993). SQ-Scores range from 0 (no fracture) to 3 (severe fracture). New fracture = SQ score is 0 at baseline and >0 at the specified end visit.
Time Frame: Baseline and Month 12
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo Daily | Risedronate Daily
Number analyzed (Participants) | 49 | 94
Participants
  At Least One New Fracture Vertebra | 8 | 28
  No New Fractured Vertebra | 40 | 60
Statistical Analysis 1: Comparison: Placebo Daily vs Risedronate Daily; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0680, Fisher Exact

26. Secondary Outcome: New Morphometric Vertebral Fracture at Month 36, ITT Population
Description: Morphometric Vertebral Fracture measured by SQ analysis of x-rays using the Genant scoring system. (Ref: Genant 1993). SQ-Scores range from 0 (no fracture) to 3 (severe fracture). New fracture = SQ score is 0 at baseline and >0 at the specified end visit.
Time Frame: Baseline and Month 36
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo Daily | Risedronate Daily
Number analyzed (Participants) | 49 | 94
Participants
  At Least One New Fracture Vertebra | 14 | 20
  No New Fractured Vertebra | 31 | 62
Statistical Analysis 1: Comparison: Placebo Daily vs Risedronate Daily; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.4121, Fisher Exact

27. Secondary Outcome: Categorization by Number of New Morphometric Vertebral Fracture at Month 12, ITT
Description: Patients with 1 or more New Morphometric Vertebral Fracture as measured by SQ analysis of x-rays using the Genant scoring system (Ref: Genant 1993). SQ-Scores range from 0 (no fracture) to 3 (severe fracture). Incidence = SQ score is 0 at baseline and >0 at post-baseline.
Time Frame: Baseline and Month 12
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo Daily | Risedronate Daily
Number analyzed (Participants) | 49 | 94
Participants
  No New Fractured Vertebra | 40 | 60
  One Fractured Vertebra | 3 | 17
  Two Fractured Vertebra | 2 | 8
  Three or more Fractured Vertebra | 3 | 3
Statistical Analysis 1: Comparison: Placebo Daily vs Risedronate Daily; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.3658, Savage Exact Test

28. Secondary Outcome: Categorization by Number of New Morphometric Vertebral Fracture at Month 36, ITT
Description: as for outcome 27
Time Frame: Baseline and Month 36
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo Daily | Risedronate Daily
Number analyzed (Participants) | 49 | 94
Participants
  No New Fractured Vertebra | 31 | 62
  One Fractured Vertebra | 6 | 10
  Two Fractured Vertebra | 5 | 7
  Three or more Fractured Vertebra | 3 | 3
Statistical Analysis 1: Comparison: Placebo Daily vs Risedronate Daily; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.3408, Savage Exact Test

29. Secondary Outcome: Incidence New Vertebral Fractures by SQ (Semi-Quantitative) Score, Patients Aged 4-9 Years, Month 12, ITT Population
Description: Patients aged 4-9 years with new morphometric vertebral fractures as measured by SQ analysis of x-rays using the Genant scoring system at Month 12 +/- 14 days. (Ref: Genant 1993). SQ Score mild - 0/no fracture to Grade 1, Moderate to Severe - change from 0/no fracture to Grade 2-3.
Time Frame: Month 12
Population: ITT Population, Number of Participants Analyzed = Number of participants with baseline and Month 12 data
Measure: Number; unit: Participants
Arm/Group | Placebo Daily | Risedronate Daily
Number analyzed (Participants) | 28 | 53
Participants
  Number Patients with New Vertebral Fractures | 7 | 19
  Number of New Vertebral Fractures | 19 | 32
  Number Patients New Fractures & Mild SQ Score | 7 | 17
  Number Patients New Fractures & Mod/Sev SQ Score | 3 | 3

30. Secondary Outcome: Incidence New Vertebral Fractures by SQ Score, Patients Aged 10-15 Years, Month 12, ITT Population
Description: Patients aged 10-15 years with new morphometric vertebral fractures as measured by SQ analysis of x-rays using the Genant scoring system at Month 12 +/- 14 days. (Ref: Genant 1993). SQ Score mild - 0/no fracture to Grade 1, Moderate to Severe - change from 0/no fracture to Grade 2-3.
Time Frame: Month 12
Population: ITT Population, Number of Participants Analyzed = Number of participants at baseline and Month 12 data
Measure: Number; unit: Participants
Arm/Group | Placebo Daily | Risedronate Daily
Number analyzed (Participants) | 21 | 41
Participants
  Number Patients with New Vertebral Fractures | 1 | 10
  Number of New Vertebral Fractures | 1 | 13
  Number Patients New Fractures & Mild SQ Score | 1 | 10
  Number Patients New Fractures & Mod/Sev SQ Score | 0 | 1

31. Secondary Outcome: Probability of Fracture in 12 Months (Kaplan-Meier Cumulative Incidence), ITT Population
Description: Long bones include radius, ulna, humerus, tibia, fibula, femur, upper limb and lower limb fracture.
Time Frame: Time to First Event (days) up to 12 Months
Population: ITT Population
Measure: Number; unit: Probability of Fractures
Arm/Group | Placebo Daily | Risedronate Daily
Number analyzed (Participants) | 49 | 94
Probability of Fractures
  Number Patients All Fractures | 24 (29) | 29
  All Fractures/Kaplan-Meier Cumulative Incidence | 0.5043 (.0740) | 0.314 (.0484)
  Number Patients Vertebral Fractures | 0 | 0
  Vertebral Fractures/Kaplan-Meier Cumulative Incid. | 0 (0) | 0 (0)
  Number Patients Non-Vertebral Fractures | 24 | 29
  Non-Vertebral Fractures/Kaplan-Meier Cum. Incid. | 0.5043 (0.0740) | 0.314 (0.0484)
  Number Patients Long Bone Non-Vertebral Fractures | 17 | 18
  Long Bone Non-Vertebral Fractures/Kaplan-Meier Cum | 0.3618 (0.0714) | 0.1954 (0.0413)
  Number Patients Other Non-Vertebral Fractures | 10 | 12
  Other Non-Vertebral Fractures/Kaplan-Meier Cum. | 0.204 (0.0576) | 0.1311 (0.0353)
Statistical Analysis 1: Comparison: Placebo Daily vs Risedronate Daily; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0253, Cox proportional hazards — All Fractures; Hazard Ratio and 95% CI based on Cox proportional hazards model stratified by age group with treatment and pooled-country as covariates; Hazard Ratio (HR) = 0.534, 95% CI [0.310 to 0.922]
Statistical Analysis 2: Comparison: Placebo Daily vs Risedronate Daily; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0253, Cox Proportional Hazard — All Non-Vertebral Fractures; [statistical method as in outcome 31, analysis 1]; Hazard Ratio (HR) = 0.534, 95% CI 2-sided [0.310 to 0.922]
Statistical Analysis 3: Comparison: Placebo Daily vs Risedronate Daily; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0501, Cox Proportional Hazards — Long Bone Non-Vertebral Fracture; [statistical method as in outcome 31, analysis 1]; Hazard Ratio (HR) = 0.487, 95% CI 2-sided [0.250 to 0.950]
Statistical Analysis 4: Comparison: Placebo Daily vs Risedronate Daily; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.2141, Cox Proportional Hazard — Other Non-Vertebral Fracture; [statistical method as in outcome 31, analysis 1]; Hazard Ratio (HR) = 0.608, 95% CI 2-sided [0.262 to 1.410]

32. Secondary Outcome: Number of Clinical Fractures, Month 12, ITT Population
Description: Long bones include radius, ulna, humerus, tibia, fibula, femur, upper limb and lower limb fracture.
Time Frame: 12 Months
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo Daily | Risedronate Daily
Number analyzed (Participants) | 49 | 94
Participants
  Number of Fractures | 38 | 42
  Number of Patients with Fractures | 24 | 29
  Number of Vertebral Fractures | 0 | 0
  Number Patients with Vertebral Fractures | 0 | 0
  Number of Non-Vertebral Fractures | 38 | 42
  Number Patients with Non-Vertebral Fractures | 24 | 29
  Number Long-Bone Non-Vertebral Fractures | 27 | 28
  Number Patients Long-Bone Non-Vertebral Fractures | 17 | 18
  Number Other Non-Vertebral Fractures | 11 | 14
  Number Patients with Other Non-Vertebral Fractures | 10 | 12
Statistical Analysis 1: Comparison: Placebo Daily vs Risedronate Daily; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0416, Wald test — All Fractures; Hazard Ratio and 95% CI based on Anderson-Gill mean intensity model stratified by age group with treatment and pooled-country as covariates; Hazard Ratio (HR) = 0.584, 95% CI [0.348 to 0.980]
Statistical Analysis 2: Comparison: Placebo Daily vs Risedronate Daily; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0416, Wald Test — Non-Vertebral Fracture; [statistical method as in outcome 32, analysis 1]; Hazard Ratio (HR) = 0.584, 95% CI 2-sided [0.348 to 0.980]
Statistical Analysis 3: Comparison: Placebo Daily vs Risedronate Daily; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0799, Wald Test — Long Bone Non-Vertebral Fracture; [statistical method as in outcome 32, analysis 1]; Hazard Ratio (HR) = 0.543, 95% CI 2-sided [0.274 to 1.076]
Statistical Analysis 4: Comparison: Placebo Daily vs Risedronate Daily; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.682, Wald Test — Other Non-Vertebral Fracture; [statistical method as in outcome 32, analysis 1]; Hazard Ratio (HR) = 0.682, 95% CI 2-sided [0.304 to 1.532]

33. Secondary Outcome: Serum BAP - Percent Change From Baseline to Month 12, ITT Population
Description: Serum Bone Alkaline Phosphatase (BAP - bone formation marker). Negative percent changes indicate response to treatment.
Time Frame: Baseline and 12 Months
Population: ITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Placebo Daily | Risedronate Daily
Number analyzed (Participants) | 49 | 94
Percent Change | 6.783 [-2.107 to 15.674] | -4.895 [-11.509 to 1.719]
Statistical Analysis 1: Comparison: Placebo Daily vs Risedronate Daily; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0318, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -11.678, 95% CI [-22.325 to -1.031]

34. Secondary Outcome: Serum BAP - Percent Change From Baseline to Month 24, ITT Population
Description: Serum Bone Alkaline Phosphatase (BAP - bone formation marker). Negative percent changes indicate response to treatment.
Time Frame: Baseline and 24 Months
Population: ITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Placebo Daily | Risedronate Daily
Number analyzed (Participants) | 49 | 94
Percent Change | -11.196 [-20.748 to -1.643] | -11.128 [-18.286 to -3.971]
Statistical Analysis 1: Comparison: Placebo Daily vs Risedronate Daily; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.9907, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.067, 95% CI 2-sided [-11.401 to 11.536]

35. Secondary Outcome: Serum BAP - Percent Change From Baseline to Month 36, ITT Population
Description: Serum Bone Alkaline Phosphatase (BAP - bone formation marker). Negative percent changes indicate response to treatment.
Time Frame: Baseline and 36 Months
Population: ITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Placebo Daily | Risedronate Daily
Number analyzed (Participants) | 49 | 94
Percent Change | -19.884 [-28.658 to -11.109] | -24.570 [-31.304 to -17.836]
Statistical Analysis 1: Comparison: Placebo Daily vs Risedronate Daily; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.3826, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -4.686, 95% CI 2-sided [-15.276 to 5.903]

36. Secondary Outcome: Urine NTX/Cr - Percent Change From Baseline at Month 12, ITT Population
Description: Urine type-I collagen N-telopeptide/creatinine (NTX/Cr; bone resorption marker). Negative percent changes indicate response to treatment.
Time Frame: Baseline and Endpoint / Month 12
Population: ITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Placebo Daily | Risedronate Daily
Number analyzed (Participants) | 49 | 94
Percent Change | -14.556 [-24.218 to -4.894] | -41.185 [-48.625 to -33.745]
Statistical Analysis 1: Comparison: Placebo Daily vs Risedronate Daily; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -26.629, 95% CI [-38.089 to -15.169]

37. Secondary Outcome: Urine NTX/Cr - Percent Change From Baseline at Month 24, ITT Population
Description: as for outcome 36
Time Frame: Baseline and Month 24
Population: ITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Placebo Daily | Risedronate Daily
Number analyzed (Participants) | 49 | 94
Percent Change | -40.358 [-54.722 to -25.994] | -31.318 [-42.478 to -20.158]
Statistical Analysis 1: Comparison: Placebo Daily vs Risedronate Daily; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.3075, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 9.040, 95% CI 2-sided [-8.433 to 26.512]

38. Secondary Outcome: Urine NTX/Cr - Percent Change From Baseline at Month 36, ITT Population
Description: as for outcome 36
Time Frame: Baseline and Month 36
Population: ITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Placebo Daily | Risedronate Daily
Number analyzed (Participants) | 49 | 94
Percent Change | -47.570 [-57.317 to -37.823] | -52.609 [-60.203 to -45.015]
Statistical Analysis 1: Comparison: Placebo Daily vs Risedronate Daily; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.3998, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -5.039, 95% CI 2-sided [-16.849 to 6.772]

39. Secondary Outcome: Wong-Baker FACES Pain Rating Scale - Change From Baseline to Month 12, ITT Population
Description: Wong-Baker FACES Pain Rating Scale (pain assessment scale using facial expressions, translated into a range from 0= no pain [smiling face] to 10= worst pain possible [distorted face with tears]; negative values indicate decrease in pain). Reference: Wong DL et al.
Time Frame: Baseline and Month 12
Population: ITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a Scale
Arm/Group | Placebo Daily | Risedronate Daily
Number analyzed (Participants) | 49 | 94
Units on a Scale | -0.056 [-0.471 to 0.358] | -0.409 [-0.712 to -0.106]
Statistical Analysis 1: Comparison: Placebo Daily vs Risedronate Daily; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.1592, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.352, 95% CI [-0.845 to 0.140]

40. Secondary Outcome: Bone Age (Years), Change From Baseline to Month 12, ITT Population
Description: Bone Age determined by visual assessment of hand / wrist radiographs.
Time Frame: Baseline and Month 12
Population: ITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Years
Arm/Group | Placebo Daily | Risedronate Daily
Number analyzed (Participants) | 49 | 94
Years | 0.956 [0.756 to 1.155] | 1.083 [0.935 to 1.231]
Statistical Analysis 1: Comparison: Placebo Daily vs Risedronate Daily; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.2917, ANOVA; LS means and p-value are from ANOVA model with fixed effects for age group, treatment and pooled center for post-baseline; Mean Difference (Net) = 0.127, 95% CI [-0.111 to 0.365]

41. Secondary Outcome: Bone Age (Years), Change From Baseline to Month 24, ITT Population
Description: Bone Age determined by visual assessment of hand / wrist radiographs.
Time Frame: Baseline and Month 24
Population: ITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Years
Arm/Group | Placebo Daily | Risedronate Daily
Number analyzed (Participants) | 49 | 94
Years | 2.147 [1.888 to 2.407] | 2.155 [1.962 to 2.347]
Statistical Analysis 1: Comparison: Placebo Daily vs Risedronate Daily; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.9622, ANOVA; LS mean and p-value are from ANOVA model adjusted by baseline and fixed effects for age group, treatment and pooled center for post-baseline; Mean Difference (Net) = 0.007, 95% CI [-0.304 to 0.319]

42. Secondary Outcome: Bone Age (Years), Change From Baseline to Month 36, ITT Population
Description: Bone Age determined by visual assessment of hand / wrist radiographs.
Time Frame: Baseline and Month 36
Population: ITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Years
Arm/Group | Placebo Daily | Risedronate Daily
Number analyzed (Participants) | 49 | 94
Years | 3.087 [2.800 to 3.374] | 3.096 [2.879 to 3.312]
Statistical Analysis 1: Comparison: Placebo Daily vs Risedronate Daily; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.9596, ANOVA; LS means and p-value are from ANOVA model adjusted by baseline and fixed effects for age group, treatment and pooled center for post-baseline; Mean Difference (Net) = 0.009, 95% CI 2-sided [-0.336 to 0.354]

43. Secondary Outcome: Annualized Growth Velocity - Change From Baseline to Month 12, ITT Population
Description: Annualized Growth Velocity [= bone age change from baseline x (365.25/time in days between baseline and the bone age measurement)]
Time Frame: Baseline and Month 12
Population: ITT Population, Number of Participants Analyzed = Number of participants at baseline and Month 12 data
Measure: Least Squares Mean (95% Confidence Interval); unit: Change in Annualized Growth Velocity
Arm/Group | Placebo Daily | Risedronate Daily
Number analyzed (Participants) | 49 | 94
Change in Annualized Growth Velocity | 0.895 [0.709 to 1.080] | 1.002 [0.865 to 1.138]
Statistical Analysis 1: Comparison: Placebo Daily vs Risedronate Daily; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.3400, ANOVA; [statistical method as in outcome 40, analysis 1]; Mean Difference (Net) = 0.107, 95% CI [-0.114 to 0.328]

44. Secondary Outcome: Annualized Growth Velocity - Change From Baseline to Month 36, ITT Population
Description: as for outcome 43
Time Frame: Baseline and Month 36
Population: ITT Population, Number of Participants Analyzed = Number of participants at baseline and Month 12 data
Measure: Least Squares Mean (95% Confidence Interval); unit: Change in Annualized Growth Velocity
Arm/Group | Placebo Daily | Risedronate Daily
Number analyzed (Participants) | 49 | 94
Change in Annualized Growth Velocity | 0.982 [0.886 to 1.077] | 1.011 [0.941 to 1.081]
Statistical Analysis 1: Comparison: Placebo Daily vs Risedronate Daily; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.6218, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.029, 95% CI 2-sided [-0.084 to 0.142]

ADVERSE EVENTS:
Time Frame: 36 months: One year double-blind treatment, 2 years open-label risedronate treatment
Groups:
- Years 2 & 3 Placebo-Risedronate: Year 1 Placebo Double-Blind, Years 2 & 3 Open-Label Risedronate
- Years 2 & 3 Risedronate: Years 1-3 Risedronate, Double-Blind Year 1, Open-Label Years 2 & 3
Arm/Group | Placebo Daily | Risedronate Daily | Years 2 & 3 Placebo-Risedronate | Years 2 & 3 Risedronate
Serious Adverse Events (participants affected / at risk) | 8/49 | 11/94 | 13/49 | 16/87
Other Adverse Events (participants affected / at risk) | 47/49 | 86/94 | 46/49 | 79/87
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Daily (N=49) | Risedronate Daily (N=94) | Years 2 & 3 Placebo-Risedronate (N=49) | Years 2 & 3 Risedronate (N=87)
Femur fracture (Injury, poisoning and procedural complications) | 7 (8) | 4 (7) | 6 (7) | 3 (5)
Forearm fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 1 (1) | 2 (2)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Ulna fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 2 (2) | 2 (3)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Mastoiditis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Humerus Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ilium Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pelvic Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rib Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cervical Vertebral Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hand Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Patella Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tympanic Membrane Perforation (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Device Failure (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Benign Bone Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Daily (N=49) | Risedronate Daily (N=94) | Years 2 & 3 Placebo-Risedronate (N=49) | Years 2 & 3 Risedronate (N=87)
Upper respiratory tract infection (Infections and infestations) | 3 (4) | 8 (13) | 4 (7) | 7 (9)
Bronchitis (Infections and infestations) | 3 (7) | 7 (13) | 2 (5) | 8 (13)
Nasopharyngitis (Infections and infestations) | 3 (3) | 7 (8) | 3 (3) | 9 (10)
Respiratory tract infection (Infections and infestations) | 1 (2) | 6 (11) | 3 (10) | 7 (16)
Influenza (Infections and infestations) | 2 (3) | 5 (6) | 2 (2) | 8 (8)
Varicella (Infections and infestations) | 0 (0) | 5 (5) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 3 (3) | 3 (7) | 2 (2) | 1 (1)
Tonsillitis (Infections and infestations) | 3 (3) | 3 (3) | 1 (1) | 3 (3)
Gastroenteritis (Infections and infestations) | 5 (5) | 1 (1) | 4 (8) | 8 (9)
Fall (Injury, poisoning and procedural complications) | 14 (21) | 19 (24) | 22 (31) | 36 (55)
Femur fracture (Injury, poisoning and procedural complications) | 8 (9) | 9 (12) | 9 (11) | 4 (7)
Joint sprain (Injury, poisoning and procedural complications) | 4 (4) | 9 (12) | 3 (6) | 6 (6)
Contusion (Injury, poisoning and procedural complications) | 3 (3) | 6 (6) | 2 (2) | 7 (10)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 6 (7) | 5 (5) | 7 (7)
Hand fracture (Injury, poisoning and procedural complications) | 3 (3) | 5 (6) | 11 (11) | 12 (17)
Tibia fracture (Injury, poisoning and procedural complications) | 2 (3) | 5 (5) | 7 (11) | 7 (7)
Joint injury (Injury, poisoning and procedural complications) | 3 (4) | 4 (4) | 4 (6) | 5 (5)
Limb injury (Injury, poisoning and procedural complications) | 3 (5) | 3 (4) | 3 (3) | 4 (8)
Ulna fracture (Injury, poisoning and procedural complications) | 4 (5) | 2 (3) | 5 (6) | 9 (12)
Muscle strain (Injury, poisoning and procedural complications) | 3 (4) | 2 (3) | 1 (1) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 4 (5) | 1 (1) | 3 (3) | 11 (11)
Wrist fracture (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 (8) | 20 (27) | 7 (7) | 11 (23)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 16 (20) | 7 (7) | 13 (20)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 9 (11) | 2 (2) | 3 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (11) | 8 (11) | 8 (11) | 5 (11)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 5 (5) | 4 (4) | 2 (3)
Vomiting (Gastrointestinal disorders) | 3 (5) | 14 (28) | 5 (13) | 5 (7)
Abdominal pain upper (Gastrointestinal disorders) | 4 (6) | 10 (10) | 6 (7) | 3 (6)
Abdominal pain (Gastrointestinal disorders) | 7 (14) | 8 (8) | 6 (6) | 5 (6)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 6 (6) | 3 (4) | 7 (7)
Nausea (Gastrointestinal disorders) | 6 (7) | 4 (4) | 4 (5) | 4 (4)
Pain (General disorders) | 5 (6) | 14 (16) | 1 (1) | 3 (5)
Pyrexia (General disorders) | 2 (2) | 8 (8) | 7 (8) | 5 (12)
Headache (Nervous system disorders) | 4 (4) | 19 (25) | 4 (5) | 8 (13)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 9 (17) | 4 (5) | 8 (18)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 5 (5) | 4 (4) | 2 (7)
Seasonal allergies (Immune system disorders) | 0 (0) | 5 (5) | 1 (2) | 3 (6)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 4 (4) | 9 (9) | 6 (9) | 12 (14)
Eye disorders (Eye disorders) | 3 (3) | 4 (6) | 3 (3) | 1 (1)
Humerus Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 3 (3) | 5 (6)
Forearm Fracture (Injury, poisoning and procedural complications) | 2 (2) | 3 (3) | 5 (6) | 3 (3)
Clavicle Fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 3 (3) | 2 (2)
Fibula Fracture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 4 (4) | 2 (2)
Dyspepsia (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 3 (3) | 2 (2)
Ear Pain (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 3 (3) | 1 (4)
Psychiatric Disorders (Psychiatric disorders) | 1 (1) | 2 (2) | 3 (3) | 2 (2)

LIMITATIONS AND CAVEATS:
The clinical meaningfulness of new fractures in the thoracic spine scored as Genant Grade I is unclear, thus the morphometric vertebral fracture data are evaluated further.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The findings of the study may be published in a scientific journal or presented at a scientific meeting. Before submitting the results of the study for publication or presentation, the Investigator will allow the Sponsor 30 days in which to review and comment on the manuscript.